CLINICAL TRIAL: NCT03411824
Title: Lung Ultrasound for Community-acquired Pneumonia Diagnosis in Emergency Medicine
Acronym: ECHOPAC
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC16_0439
Record Dates: First submitted 2017-11-30; First posted 2018-01-26 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Community Acquired Pneumonia
Keywords: diagnosis; Point-of-Care-Ultrasound; lung ultrasound
MeSH Terms: conditions — Community-Acquired Pneumonia; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — Non applicable

SUMMARY:
Community-acquired pneumonia (CAP) is frequently suspected in the Emergency Department (ED). However, usual diagnosis procedure based on clinical features and chest X-Ray has rather bad performances.

A recent study on CT performance in suspected CAP found that 58% of classifications were modified by CT when compared with usual procedure. However, extended CT usage in CAP diagnosis is associated with many limitations :

availability in a majority of ED, delay, cost and irradiation, in particular In young patients.

Lung Ultrasound (LUS) has good performances in CAP diagnosis even when compared with CT. It is a rapid, inexpensive, radiation-free tool available in a majority of ED. It is performed at the patient's bedside with immediate results. The learning curve allows Emergency Physicians (EP) to perform this exam after a relative brief training.

The Investigators aim to investigate LUS performances in clinically suspected CAP authentication , and assesses specific diagnostic contributions and impact on antibiotic prescriptions .

DETAILED DESCRIPTION:
120 patients will be enrolled on CAP suspicion. All explorations (radiography…) and biological exams (blood culture…) will be performed as usual to build physician primary diagnosis. Complementarily, an EP will be realized and final diagnosis will be made by physician. Finally, at Day28 expert adjudication committee will authentic diagnosis considering explorations and clinical issues. Frequency of discordant diagnosis between 1st and 2nd assessment and against expert will be measured Primary Purpose: diagnostic Study Phase: Not Applicable Intervention Model: NA Number of Arms: 1 Masking: open label, Masked Roles: NA Allocation: NA Study Endpoint Classification: efficacy Enrollment: 120 subjects (anticipated )

ELIGIBILITY:
Inclusion Criteria :

- clinical suspicion of PAC

Exclusion Criteria :

* documented end-of-life
* pregnancy
* seriously ill patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 120 patients will be enrolled on CAP suspicion. All explorations (radiography…) and biological exams (blood culture…) will be performed as usual to build physician primary diagnosis. Complementarily, an EP will be realized and final diagnosis will be made by physician. Finally, at Day28 expert adjudication committee will authentify diagnosis considering explorations and clinical issues. Frequency of discordant diagnosis between 1st and 2nd assessment and against expert will be measured
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2016-11-08 (Actual); Primary Completion 2019-02-08 (Actual); Study Completion 2019-02-08 (Actual)

PRIMARY OUTCOMES:
Frequency of PAC classification modification (definite, probable, possible, excluded) after LUS realization | Day 0
  95% confidence interval of CAP classification modification frequency before and after LUS realization

SECONDARY OUTCOMES:
Concordancy of CAP classification diagnosis concordancy ( after LUS) compared to adjudication committee | 28 days after enrollment
  CAP classification (definite, probable, possible, excluded) and kappa coefficient.
Frequency of Antibiotic prescription modification after LUS | Day 0
  95% confidence interval of antibiotic prescription intention frequency

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Le Conte, Pr, Principal Investigator — Nantes University Hospital
Locations (4):
- France (4):
  - La Roche Sur Yon Hospital, La Roche-sur-Yon
  - Nantes University Hospital, Nantes
  - Poitiers University Hospital, Poitiers
  - Saint-Nazaire Hospital, Saint-Nazaire

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Javaudin F, Marjanovic N, de Carvalho H, Gaborit B, Le Bastard Q, Boucher E, Haroche D, Montassier E, Le Conte P. Contribution of lung ultrasound in diagnosis of community-acquired pneumonia in the emergency department: a prospective multicentre study. BMJ Open. 2021 Sep 24;11(9):e046849. doi: 10.1136/bmjopen-2020-046849. PMID 34561254